CLINICAL TRIAL: NCT05387577
Title: Coagulation Activation and Fibrinolysis With Sublingual Versus Oral Versus Transdermal Estradiol in Transgender Women
Brief Title: Coagulation and Fibrinolysis of Estradiol in Transwomen
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: per MCW IRB
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jenna Sarvaideo, Assistant Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRO00036346
Record Dates: First submitted 2022-04-16; First posted 2022-05-24 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Transgenderism; Clotting Disorder
Keywords: Estradiol; Estrogens; Hormones; Hormones, Hormone Substitutes, Hormone Antagonists; Physiological Effects of Drugs; Transgender
MeSH Terms: conditions — Transsexualism; Hemostatic Disorders | interventions — Estradiol; Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sublingual Estradiol (Active Comparator): Sublingual estradiol administered for 8 weeks
  Interventions: Drug: Estradiol Tablets
- Oral Estradiol (Active Comparator): Oral estradiol administered for 8 weeks
  Interventions: Drug: Estradiol Tablets
- Transdermal Estradiol (Active Comparator): Transdermal estradiol administered for 8 weeks
  Interventions: Drug: Transdermal patch

INTERVENTIONS:
Drug: Estradiol Tablets — Oral estradiol will be taken sublingually, 1 mg BID for 8 weeks
  Other Names: Sublingual estradiol tablets
  Arms: Sublingual Estradiol
Drug: Transdermal patch — Estradiol patch therapy for 8 weeks
  Other Names: Transdermal estradiol patch
  Arms: Transdermal Estradiol
Drug: Estradiol Tablets — Oral estradiol 1 mg BID for 8 weeks
  Other Names: Oral Estradiol tablets
  Arms: Oral Estradiol

SUMMARY:
The specific aim for our study is to measure coagulation system activation and fibrinolysis following transdermal versus sublingual versus oral estradiol versus in transgender women.

Hypothesis: Transdermal estradiol will result in less coagulation system activation and no effect on plasminogen activator inhibitor (PAI-1) or tissue-type plasminogen activator (t-PA). Oral estradiol will result in the most coagulation system activation and effect on PAI-1 and t-PA: Oral estradiol > sublingual estradiol > transdermal estradiol.

A prospective crossover study will include ten subjects given estradiol 1 mg daily and instructed to take it orally, sublingually, or transdermal for 2 months with a 2-week washout period between routes of administration. Labs will be measured 7 times during the study.

DETAILED DESCRIPTION:
Subjects will report to our Adult Translational Research Unit for labs at baseline (2 weeks after HRT washout if needed). Both fibrinolysis and testosterone labs have a diurnal variation. Therefore, fasting labs will be drawn at approximately 8 AM. Five subjects will start oral estradiol and 5 will start sublingual estradiol for 8 weeks. Froedtert's Pharmacy Investigational Drug Service will provide the study estradiol. There will be a 2-week washout period between treatment periods. Fasting labs will be drawn at approximately 8 AM prior to Treatment Period 2. The groups will switch therapy. Those that took oral estradiol during Treatment Period 1 will take sublingual estradiol for 8 weeks. Those that took sublingual estradiol during Treatment Period 1 will take oral estradiol for 8 weeks. Finally, all subjects will start the transdermal for 8 weeks for Treatment Period 3. Final set of labs will be drawn at approximately 8 AM 2 weeks after Treatment Period 3. The investigators will call subjects every 2 weeks to assess their adherence to the treatment protocol and remind them of the importance of allowing the tablet to dissolve when taking estradiol sublingually.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Gender identity of male to female or transwoman

Exclusion Criteria:

* Liver disease
* History of blood clot
* Bleeding disorder
* Active or recent (e.g., within the past year) stroke
* Myocardial infarction,
* History of orchiectomy
* History of breast cancer,
* Known sensitivity or allergy to any components of the medications used
* Currently taking a potent CYP3A4 inhibitor or inducer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transwoman (gender identity female, assigned male at birth)
Enrollment: 6 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Coagulation system activation and fibrinolysis due to estradiol administration | 8 months
  Comparison of morning fasting labs (fibrinogen, von-Willebrand Factor (vWF) ristocetin cofactor, vWF antigen, D-dimer, protein C activity, free protein S activity, Factors VII, VIII, IX, thrombin generation, plasminogen activator inhibitor (PAI-1), tissue-type plasminogen activator (t-PA) and t-PA activity) in transgender women taking estradiol via different routes of administration. Our hypothesis is that transdermal estradiol will result in less coagulation system activation and no effect on PAI-1 or t-PA. Oral estradiol will result in the most coagulation system activation and will effect PAI-1 and t-PA: Oral estradiol > sublingual estradiol > transdermal estradiol.

SECONDARY OUTCOMES:
Thrombotic risk due to estradiol administration | 8 months
  Thrombotic risk will be assessed in transgender women by measuring estrone and thrombin generation and comparing them between the different routes of estradiol administration (transdermal versus sublingual versus oral).

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Sarvaideo, DO, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 3 months after publication
Access Criteria: IPD will be shared if PI is directly contacted and asked for the above information.